CLINICAL TRIAL: NCT06471777
Title: Proactive Prescription-based Fluid Management Versus Usual Care in Critically Ill Patients on Kidney Replacement Therapy Trial in UK
Brief Title: Prescription-based Fluid Management Versus Usual Care in Critically Ill Patients on KRT Trial in UK
Acronym: PROBE Fluid UK
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: Université de Montréal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GSTT V1
Record Dates: First submitted 2024-06-18; First posted 2024-06-24 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Acute Renal Failure on Dialysis (Disorder)
Keywords: acute kidney injury; dialysis; fluid removal
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Protocol-based fluid removal (Experimental): The intervention will consist of 3 components:
  The first component of this prescription will be to define the 24h-fluid balance target. The second component is to specify a prescription for fluid removal. The third component is to prompt a daily re-evaluation of fluid intake and fluid balance by the attending care team.
  Interventions: Procedure: Fluid removal
- Usual care (No Intervention): Fluid removal during KRT will be determined by the attending clinical team.

INTERVENTIONS:
Procedure: Fluid removal — Fluid removal during kidney replacement therapy
  Arms: Protocol-based fluid removal

SUMMARY:
The PROBE Fluid UK randomised controlled trial compares a protocol-based fluid removal strategy with usual care in critically ill patients with acute kidney injury receiving kidney replacement therapy.

DETAILED DESCRIPTION:
Severe acute kidney injury (AKI) in the intensive care unit (ICU) is almost uniformly complicated by fluid accumulation, often leading to fluid overload. Congestion resulting from fluid accumulation is believed to contribute to organ failure. Removal of excess fluid is a central component of dialysis treatment, also known as kidney replacement therapy (KRT). However, there remain important knowledge gaps in our ability to remove excess fluid effectively and safely. If fluid is removed too slowly, fluid overload and its complications persist for longer. If fluid is removed too fast during KRT, patient's blood pressure may drop (ie hemodynamic instability may occur) which may precipitate complications.

The optimal fluid management strategy is currently unknown.

The PROBE Fluid UK study is a randomized clinical trial comparing a protocol-based fluid removal strategy with usual care in critically ill patients with AKI receiving KRT. The fluid management protocol is intended to achieve neutral or negative daily fluid balance by both preventing and treating fluid accumulation.

The primary objective of this trial is to determine whether the intervention results in a difference in cumulative fluid balance from day of randomization to 5 days later. Secondary outcomes will include short-term patient outcomes, safety outcomes, and health resource utilization related to KRT delivery.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients aged ≥18 years
2. Admitted to the intensive care unit
3. Acute kidney injury defined by the KDIGO criteria
4. Planned initiation of KRT within 12 hours or the receipt of KRT for AKI for ≤48 hours

Exclusion Criteria:

1. Lack of commitment to maintain kidney, pharmacologic or respiratory support at the time of screening, or probable transition to comfort care within 48 hours according to the treating clinician
2. Probable discharge from the ICU within 48 hours according to treating clinician
3. Severe burn injury (>10% of body surface area)
4. Severe abnormality in serum sodium (>155 or <120 mmol/L)
5. Important ongoing fluid losses are present and/or are expected to require continued maintenance IV fluids during the next 48 hours
6. The clinical care team believes that the proposed intervention is inappropriate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
fluid balance | day 5 after randomization
  cumulative fluid balance

SECONDARY OUTCOMES:
enrolment | 20 months
  Proportion of eligible patients who were enrol in the trial
mortality | 90 days after randomization
  all-cause mortality
ICU stay | 90 days after randomization
  Number of ICU free days
vasoactive therapy | 28 days after randomization
  Number of vasoactive therapy-free days
mechanical ventilation | 28 days after randomization
  Number of mechanical ventilation-free days
KRT duration | 5 days
  hours of KRT support

IPD SHARING:
Plan to Share IPD: No